CLINICAL TRIAL: NCT05786703
Title: Integrated Hypertension and Diabetes Mellitus Type II Treatment and Care Among People Living With HIV/AIDS Attending Care and Treatment Center in Dar es Salaam, Tanzania
Brief Title: Integrated Hypertension and Diabetes Mellitus Type II Treatment and Care Among People Living With HIV/AIDS
Status: Completed | Type: Observational
Sponsor: Muhimbili University of Health and Allied Sciences (Other)
Responsible Party: Principal Investigator, Atuganile Musyani, Principal Investigator, Muhimbili University of Health and Allied Sciences
Other Study IDs: MUHAS-REC-1-2020-074
Record Dates: First submitted 2023-03-12; First posted 2023-03-27 (Actual); Last update posted 2023-05-08 (Actual); Status verified 2023-05

CONDITIONS: Diabetes Mellitus; Hypertension; HIV Infections
MeSH Terms: conditions — Diabetes Mellitus; Hypertension; HIV Infections | interventions — Blood Pressure

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Biochemical, weight measurements, Blood pressure and blood sugar level — At first visit short interview using the STEPwise approach of the STEPS surveillance tool for NCDs from the WHO will be conducted. On subsequent visits, hypertension and blood sugar level and cholesterol levels will be measured and adherence to medication will be assessed. The patient's registry will be developed following recommendation from the HEARTS technical package of World Health Organization (WHO) with some modification if needed.

SUMMARY:
This project was a facility-based program intervention for People Living with HIV (PLHIV) aged 18 years and above who attended a Care and Treatment Center (CTC) in Dar es Salaam, Tanzania. Clients received preventive, diagnostic, and treatment services for Hypertension (HTN) and Type Two Diabetes Mellitus (T2DM). The primary health outcomes were all-cause mortality, disease-specific morbidity, HTN, and T2DM control rates. Secondary outcomes included access to care, retention in care adherence, and quality of care. Results obtained can be used to strengthen Non-Communicable Diseases (NCDs) care delivery in HIV/AIDS care in CTC in Tanzania.

DETAILED DESCRIPTION:
A cohort of patients who were diagnosed with hypertension and diabetes was created and followed up for 6 months. Patients were required to attend clinics on a monthly basis. At the first visit short interview using the STEPwise approach of the STEPS surveillance tool for NCDs from the World Health Organization (WHO) was conducted. On subsequent visits, hypertension and blood sugar levels and cholesterol levels will be measured and adherence to medication were assessed. The patient registry was developed following recommendations from the HEARTS (Healthy lifestyle, Evidence-based protocols, Access to essential medicines and technology, Risk-based Cardiovascular Disease (CVD) management, Team-based care Guidance Systems for monitoring)technical package of WHO with some modifications if needed. A simple surveillance system was developed for all patients diagnosed with hypertension and diabetes so that there is continuous evaluation and monitoring of all patients attending NCDs care at the HIV clinic.

ELIGIBILITY:
Inclusion Criteria:

All PLHIV who attended CTC 18 years and above

Exclusion Criteria:

* Pregnant women living with HIV/AIDS
* Patients with mental diseases.

Ages: 18 Years to 54 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The target population was PLHIV aged 18 years or above attending Temeke RRH in Temeke District in Dar es Salaam, Tanzania. We used convinient sampling to select PLHIV who attended CTC within the 5 days of data collection. Clients were randomly selected based on availability at the time of interview. The project excluded pregnant women living with HIV/AIDS and patients with mental diseases.
Sampling Method: Non-Probability Sample
Enrollment: 333 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2020-06-30 (Actual)

PRIMARY OUTCOMES:
CHANGE IN BLOOD PRESSURE LEVEL | SIX MONTHS
  Change in the mean blood pressure at the beginning and the end of the study

CONTACTS AND LOCATIONS:
Overall Officials: Atuganile Musyani, Masters, Principal Investigator — Muhimbili University of Health and Allied Sciences
Locations (1):
- Temeke Regional Referral Hospital, Dar es Salaam, Tanzania